CLINICAL TRIAL: NCT01013818
Title: A Phase 1, Multi-Center, Open-Label, Dose Escalation Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of HGS1029 in Subjects With Relapsed or Refractory Lymphoid Malignancies
Brief Title: A Study of HGS1029 in Subjects With Relapsed or Refractory Lymphoid Malignancies
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to slow accrual
Sponsor: Human Genome Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGS1029-C1080
Record Dates: First submitted 2009-11-03; First posted 2009-11-16 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2013-08

CONDITIONS: Lymphoid Malignancies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HGS1029 (Experimental)
  Interventions: Drug: HGS1029

INTERVENTIONS:
Drug: HGS1029 — HGS1029 will be given as a 15-minute IV infusion (in the vein) once weekly for 3 consecutive weeks, followed by 1 week off.

SUMMARY:
The purpose of this study is to determine if HGS1029 is safe and well tolerated in patients with relapsed or refractory lymphoid malignancies.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed relapsed/refractory lymphoid malignancies
* Previously treated with at least 2 therapeutic regimens
* ECOG performance < 2.
* Life expectancy of at least 3 months
* Adequate renal function
* Adequate hematologic status
* Adequate liver function
* Transfusion independent

Exclusion Criteria:

* Received other therapy (biological or drug) to treat cancer within 4 weeks prior to starting treatment with HGS1029 or who exhibit persistent clinical evidence of cancer treatment toxicity
* The use of systemic corticosteroids within 1 week of starting treatment with HGS1029
* Evidence of active bacterial, viral or fungal infection within 2 weeks before starting treatment with HGS1029
* Known HIV infection
* Positive for hepatitis B surface antigen or positive hepatitis C antibody
* Grade 2 or greater neuropathy
* Pregnant female or nursing mother
* Males or females who do not agree to use effective contraception during the study and through at least 30 days after the last dose of HGS1029

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2009-10; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Type, frequency and severity of adverse events | 1 year

SECONDARY OUTCOMES:
Measure pharmacokinetic profile | 1st two months of the study
Evaluation of pharmacodynamics | 1st two months of the study
Evaluation of possible anti-tumor activity | Every 2 months while on study

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- United States (2):
  - Mayo Clinic, Rochester, Minnesota
  - Hackensack University Medical Center, Hackensack, New Jersey
- United Kingdom (3):
  - Oxford Cancer and Haematology Centre, Headington, Oxford
  - The Institute of Cancer Research, Belmont, Sutton, Surrey
  - Cancer Research UK Centre, Southampton